CLINICAL TRIAL: NCT02788422
Title: The Effectiveness of Video Discharge Instructions for Acute Otitis Media on Knowledge Acquisition and Clinical Outcomes: a Randomized Controlled Trial
Brief Title: Video Discharge Instructions for Acute Otitis Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10012437
Record Dates: First submitted 2016-05-24; First posted 2016-06-02 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (Experimental): Video discharge instructions developed using Easy Sketch Pro3TM software (Easy Sketch Pro, United Kingdom). It was created by the primary and co-investigator based results on a focus group consisting of two paediatric residents, two paediatric emergency medicine fellows, a paediatric emergency medicine nurse, and a paediatric emergency medicine staff physician.
  Interventions: Other: Video discharge instructions
- Standard of care (Active Comparator): This is a one-page paper handout created by the primary and co-investigator based results on a focus group consisting of two paediatric residents, two paediatric emergency medicine fellows, a paediatric emergency medicine nurse, and a paediatric emergency medicine staff physician.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Video discharge instructions — Online video containing information on how to manage symptoms of acute otitis media and when to return to a health care professional.
  Arms: Video
Other: Standard of Care — One page paper handout containing information on how to manage symptoms of acute otitis media and when to return to a health care professional.
  Arms: Standard of care

SUMMARY:
Thorough, understandable discharge instructions empower caregivers, allowing them to provide optimum care of their children during illness. Unfortunately discharge instructions are often incomplete and difficult to understand. The use of video discharge instructions has been shown to increase patient understanding of their illness. The investigators would like to know if using video discharge instructions for caregivers of children with middle ear infections helps to better understand how to take care of children at home, potentially allowing the child to feel better faster. The investigators will be comparing video discharge instructions to a paper handout to see if the former leads to improved well-being of the child and improved caregiver knowledge, satisfaction and anxiety.

DETAILED DESCRIPTION:
Providing patients with understandable, comprehensive discharge instructions improves compliance, thereby reducing symptoms and the functional impact of illness. Comprehensive discharge instructions also reduce patient anxiety and increases satisfaction. Unfortunately, in a busy emergency department (ED), discharge instructions are often incomplete. Furthermore, even when discharge instructions have been provided, patients often have difficulty comprehending and/or recalling them. Inadequate discharge instructions are linked to medication errors, suboptimal care post-discharge, and unnecessary return visits to the ED. Patient dissatisfaction with discharge instructions and anxiety have also been linked to poor medication compliance, and an increase in return visits.

Studies have demonstrated that knowledge of pediatric medical conditions can be enhanced through the use of video technology. Specifically, it has been shown that when video discharge instructions are used in place of, or to complement written discharge instructions, patients have a better understanding of their illness and report higher rates of satisfaction. However, no studies to date have explored if clinically relevant outcomes such as symptomatology, function and recidivism can be improved.

This study will examine the utility of video discharge instructions for the diagnosis of acute otitis media (AOM), a leading cause of health care visits among children. AOM affects up to 75% of children before school-age and is the most common illness for which antibiotics are prescribed to children in the United States. In Canada, AOM is associated with substantial use of health services (3.1 hours in an emergency department and 1.8 hours in an outpatient clinic on average per visit) and significantly burdens caregivers in the form of time spent on medical consultations, and time taken off from work. An American study estimated that the cost of one episode of AOM in a 3-month period following diagnosis was $1330.58, with the majority of that cost stemming from the indirect costs of illness, 90% of which was accrued primarily by parental time off work. In Quebec, the total annual cost to the health care system for otitis media and placement of tympanostomy tubes is more than $10 million dollars.

Pain is often substantial in the early course of AOM. Poorly controlled pain is associated with suffering and can be emotionally traumatic, causing anxiety for patients and their caregivers. Efficacious treatment for child pain is paramount in preventing protracted sensitivity to pain. Despite the magnitude of effects that acute pain can have on a child, it is often inadequately assessed and treated. In children less than two years of age, 30% of children continue to experience pain, fever, or both for up to 7 into the illness, thus highlighting the importance of caregiver education on symptom management.

Recurrent AOM is common, 5-15% of children under the age of 2 experience four or more episodes per year. Caregivers of children with recurrent AOM not only judge their child's quality of life markedly lower than caregivers of children of a general population, but also lower than those of children with mild-to-moderately severe chronic conditions. Although uncommon, AOM also has the potential to cause serious complications such as, mastoiditis and bacterial meningitis, if not treated and monitored appropriately.

The investigators hypothesize that video discharge instructions directed at caregivers of children with AOM will be associated with improved symptomatology and functional outcomes, along with improved caregiver knowledge, satisfaction, and anxiety compared to the standard of care, paper-based discharge instructions.

ELIGIBILITY:
Inclusion Criteria:

* All primary caregivers of children aged 6 months to 17 years presenting to the Emergency Department of the Children's Hospital, London Health Sciences Centre, London, Ontario
* Clinical diagnosis of AOM in the context of an upper respiratory tract infection as determined by the treating emergency physician (staff physician or fellow). The treating physician will be asked to rate, using a 10 mm visual analog scale, the likelihood that the patient has AOM using previously published diagnostic criteria. - Physician reports being at least 50% certain, on a visual analog scale in the diagnosis of AOM.

Exclusion Criteria:

* Caregivers whose children have other diagnoses (pneumonia, urinary tract infection, gastroenteritis, or any other condition requiring antibiotics or admission to hospital)
* Previous diagnosis of AOM within 7 days
* Tympanostomy tubes
* Acute tympanic membrane perforation
* Attending caregiver who is not the primary care provider
* Poor English fluency
* Lack of at least a grade 8 literacy level
* No Internet access
* No telephone access for 72 hours following discharge

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-03-17 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Daily self-reported Acute Otitis Media Symptom Severity Score | 72 hours
  At 72 hours

SECONDARY OUTCOMES:
Self-report State Trait Anxiety Inventory at discharge | 72 hours
Caregiver Satisfaction at 72 hours | 72 hours
Self-reported number of days of school/work/daycare missed at 72 hours | 72 hours
Self-reported medication administered daily for 72 hours | 72 hours
  Number of doses and type of medication administered based on self-report
Self-reported return visits to a health care provider at 72 hours | 72 hours
  Number of visits and type of health care provider and reason based on self-report
Number of times online video was viewed in 72 hours | 72 hours
Change in knowledge score on novel questionnaire before and after intervention in ED | 30 minutes
  Difference in knowledge questionnaire scores before and immediately following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Poonai, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belisle S, Dobrin A, Elsie S, Ali S, Brahmbhatt S, Kumar K, Jasani H, Miller M, Ferlisi F, Poonai N. Video Discharge Instructions for Acute Otitis Media in Children: A Randomized Controlled Open-label Trial. Acad Emerg Med. 2019 Dec;26(12):1326-1335. doi: 10.1111/acem.13839. Epub 2019 Nov 19. PMID 31742809